CLINICAL TRIAL: NCT01335945
Title: Percutaneous Cryoablation for the Palliation of Abdominal Pain Associated With Pancreatic Cancer
Brief Title: Safety and Efficacy of Cryoablation for Abdominal Pain Associated With Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment & subjects didn't survive to study end due to cancer progression.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CUC10-PAN09
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Pain; Pancreatic Cancer
Keywords: Cryoablation; Cryotherapy; Cryosurgery; Pancreas; Pancreatic Cancer; Celiac Plexus; Pain; Abdominal pain
MeSH Terms: conditions — Pain; Pancreatic Neoplasms; Abdominal Pain | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation (Other): Freezing of the celiac plexus
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — All subjects will receive cryoablation of the celiac plexus with Galil Medical cryoablation systems and needles under imaging guidance.
  Other Names: Cryotherapy; Visual-ICE cryoablation system; SeedNet cryoablation system; PresIce cryoablation system; IceRod cryoablation needles; IceRod PLUS cryoablation needles; IceRod CX cryoablation needles; IceEDGE 2.4 cryoablation needles; IceSphere cryoablation needles; IceSeed cryoablation needles

SUMMARY:
CUC10-PAN09 will evaluate the safety and efficacy of cryoablation therapy on the relief of epigastric/abdominal pain associated with pancreatic cancer.

DETAILED DESCRIPTION:
CUC10-PAN09 is a Supportive Care, Phase 1 multicenter, prospective, single arm study with subjects serving as their own control. This study is to enroll patients who will undergo cryoablation of the Celiac Plexus. Subjects will be followed for 3 months post their cryoablation procedure.

Cryoablation is the process of destroying tissue by the application of extremely cold temperatures. Galil Medical Cryoablation Systems are used as a surgical tool in the fields of general surgery, dermatology (skin), neurology (nerves), chest surgery (including lung), Ears-Nose-Throat (ENT), gynecology, oncology (cancer), proctology (colon/rectal) and urology (kidney).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years old
* Subject has unresectable or inoperable pancreatic carcinoma as determined by CT or MRI
* Subject's epigastric/abdominal 'worst pain' in the last 24 hours must be reported to be 4 or above on a scale of 0 (no pain) to 10 (pain as bad as subject can imagine) on the BPI despite pharmaceutical pain management
* ECOG of 0-3
* Platelet count >50,000
* INR <1.5

Exclusion Criteria:

* Subject's life expectancy is <3 months
* Subject has current neutropenia (ANC <1000)
* Subject unable to undergo CT or MRI
* Subject had previous ETOH neurolytic block for pancreatic cancer-related pain less than 2 weeks from screening
* Subject had surgery <4 weeks from screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Abdominal pain reduction following cryoablation of the celiac plexus | 3 Months
  Measured by the average difference of pre- and post-treatment worst pain in the last 24 hours (baseline), within 24 hours of the cryoablation procedure, 1 week, 4 weeks, 8 weeks and 12 weeks as measured on the numeric 0-10 Brief Pain Inventory (BPI) Scale

SECONDARY OUTCOMES:
Duration of abdominal pain relief | 3 Months
  Measured from the cryoablation procedure to the return of the abdominal pain
Cryoablation Procedure Information | During the procedure on the procedure day (an expected average of 3 hours)
  Number of cryoablation needles used, freeze and thaw cycles and times, method of thaw and ice formation
Hospital Duration | Participants will be followed for the duration of hospital stay, an expected average of 1 day
  Date and time of admission and discharge
Difference in average pain scores | 3 Months
  Measured from baseline to within 24 hours of the cryoablation procedure, 1 week, 4 weeks, 8 weeks and 12 weeks as measured on the numeric 0-10 Brief Pain Inventory Scale
Percentage of subjects able to reduce analgesic medications | 3 Months
  Measured from baseline to within 24 hours of the cryoablation procedure, 4, 8 and 12 weeks post cryoablation procedure
Time to maximal epigastric/abdominal pain relief after cryoablation | 3 Months
  The safety endpoint for this study is to assess the incidence and severity of intra-operative events, post operative adverse events, serious adverse events and unanticipated adverse device effects related to the cryoablation procedure
Time to recurrence of epigastric/abdominal worst pain at or above baseline | 3 Months
  Measured worst pain score in the 12 week follow-up period as measured on a numeric 0-10 Brief Pain Inventory Scale
Subject satisfaction with the amount of epigastric/abdominal pain relief from cryoablation procedure | 3 Months
  Subjects will answer questions regarding their satisfaction.
Safety assessment | 30 Days post cryoablation
  The safety endpoint for this study is to assess the incidence and severity of intra-operative events, post operative adverse events, serious adverse events and unanticipated adverse device effects related to the cryoablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: David D Childs, MD, Principal Investigator
Locations (3):
- United States (3):
  - Karmanos Cancer Institute, Detroit, Michigan
  - The Research Foundation of State University New York, Stony Brook, New York
  - University Hospitals, Cleveland, Ohio

REFERENCES:
- [Background] Xiong LL, Hwang JH, Huang XB, Yao SS, He CJ, Ge XH, Ge HY, Wang XF. Early clinical experience using high intensity focused ultrasound for palliation of inoperable pancreatic cancer. JOP. 2009 Mar 9;10(2):123-9. PMID 19287104
- [Background] Michaels AJ, Draganov PV. Endoscopic ultrasonography guided celiac plexus neurolysis and celiac plexus block in the management of pain due to pancreatic cancer and chronic pancreatitis. World J Gastroenterol. 2007 Jul 14;13(26):3575-80. doi: 10.3748/wjg.v13.i26.3575. PMID 17659707
- [Background] Kruse EJ. Palliation in pancreatic cancer. Surg Clin North Am. 2010 Apr;90(2):355-64. doi: 10.1016/j.suc.2009.12.004. PMID 20362791
- [Background] Patiutko IuI, Barkanov AI, Kholikov TK, Lagoshnyi AT, Li LI, Samoilenko VM, Afrikian MN, Savel'eva EV. [The combined treatment of locally disseminated pancreatic cancer using cryosurgery]. Vopr Onkol. 1991;37(6):695-700. Russian. PMID 1843146
- [Background] Kovach SJ, Hendrickson RJ, Cappadona CR, Schmidt CM, Groen K, Koniaris LG, Sitzmann JV. Cryoablation of unresectable pancreatic cancer. Surgery. 2002 Apr;131(4):463-4. doi: 10.1067/msy.2002.121231. PMID 11935137
- [Background] Wong GY, Schroeder DR, Carns PE, Wilson JL, Martin DP, Kinney MO, Mantilla CB, Warner DO. Effect of neurolytic celiac plexus block on pain relief, quality of life, and survival in patients with unresectable pancreatic cancer: a randomized controlled trial. JAMA. 2004 Mar 3;291(9):1092-9. doi: 10.1001/jama.291.9.1092. PMID 14996778
- [Background] Yan BM, Myers RP. Neurolytic celiac plexus block for pain control in unresectable pancreatic cancer. Am J Gastroenterol. 2007 Feb;102(2):430-8. doi: 10.1111/j.1572-0241.2006.00967.x. Epub 2006 Nov 13. PMID 17100960
- [Background] Stefaniak T, Basinski A, Vingerhoets A, Makarewicz W, Connor S, Kaska L, Stanek A, Kwiecinska B, Lachinski AJ, Sledzinski Z. A comparison of two invasive techniques in the management of intractable pain due to inoperable pancreatic cancer: neurolytic celiac plexus block and videothoracoscopic splanchnicectomy. Eur J Surg Oncol. 2005 Sep;31(7):768-73. doi: 10.1016/j.ejso.2005.03.012. PMID 15923103